CLINICAL TRIAL: NCT03901560
Title: The Effect of Music Therapy on Pediatric Patients Admitted to the Hospital for Sickle Cell or Pain Crisis
Brief Title: Music Therapy: Sickle Cell and Pain Crisis
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Collaborators: The Children's Hospital at OU Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 5897
Record Dates: First submitted 2019-04-02; First posted 2019-04-03 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Sickle Cell Crisis; Functional Abdominal Pain; Patients Followed by the Pain Team
MeSH Terms: conditions — Vaso-Occlusive Crises | interventions — Music Therapy

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Music Therapy

SUMMARY:
This study will assess whether participants who receive music therapy during inpatient care report a decrease in pain and whether music therapy influences factors such as family satisfaction.

DETAILED DESCRIPTION:
The purpose of this study is to determine if music therapy services can serve as a viable, necessary, and beneficial aspect of inpatient pain management, distraction, and coping for pediatric patients in the acute care hospital setting. The investigator will note the effect of music therapy services in conjunction with pain scores reported by the participant and an increase in self and family reported coping skills during hospitalization.

Participants will be referred by providers from pain management service, oncology/hematology service, or the gastrointestinal (GI) service for functional and abdominal pain. Participants who meet the criteria for inclusion will be selected. The study will be explained to parents and a consent form will be left for the family to review and sign at their convenience. Participants will provide a pain scale level and vitals before completing the music therapy intervention. Once the music therapy intervention is completed, the pain scale and vitals will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* 5-17 years of age
* Admitted for sickle cell crisis, functional abdominal pain, or whom the pediatric pain management team is following.

Exclusion Criteria:

* Non-English speaking
* Under 5 years old and over 17 years old
* Patients who are unable to hear or have a hearing disability
* Developmentally unable to self-report pain levels

Ages: 5 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Patients between the ages of 5-17 who either have sickle cell, are on the pain team, or functional abdominal pain
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2017-07-13 (Actual); Study Completion 2017-07-13 (Actual)

PRIMARY OUTCOMES:
How does music therapy affect perceived pain in hospitalized pediatric patients? | 30 minutes
  Do pediatric patients who receive music therapy report a decrease in pain after receiving a music therapy intervention as measured by the Wong Baker Faces Scale? The Wong Baker Faces Scale uses six different faces to assist child patients in rating their pain on a scale of '0' for no pain to '10' for severe to extreme pain.
How does music therapy influence factors such as family satisfaction and length of stay at the time of discharge? | 30 minutes
  Will music therapy result in patient and/or family satisfaction as measured by a survey administered immediately after the intervention?

IPD SHARING:
Plan to Share IPD: Undecided